CLINICAL TRIAL: NCT02602587
Title: Study of Dendrogenin A / Oxysterols Balance Between Healthy Volunteers and Acute Myeloid Leukemia Patients. Modulations of the Balance During Cytarabine/Anthracycline Treatment - OxyLAM
Brief Title: Study of Dendrogenin A / Oxysterols Balance Between Healthy Volunteers and Acute Myeloid Leukemia Patients
Acronym: OXYLAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14 7166 03
Record Dates: First submitted 2015-11-02; First posted 2015-11-11 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; Dendrogenin A; 5,6-cholesterol epoxide; 6-oxo-cholestane-3beta; 5alpha-diol; cholesterol epoxide hydrolase; oxysterols
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- blood samples and bone marrow samples (Experimental): The patients included in this study will be processed according to the standard treatment in force for their disease. This study does not in any way interfere with this treatment regimen, and is only based on additional samples of blood and bone marrow in acts planned in the prognostic or follow-up protocols. Treatment shall start within the 15 days following inclusion and first sampling.
  Interventions: Biological: Blood sample; Biological: Bone marrow sample

INTERVENTIONS:
Biological: Blood sample — additional samples of blood in acts planned in the prognostic or follow-up protocols.
Biological: Bone marrow sample — additional bone marrow sample in acts planned in the prognostic or follow-up protocols.

SUMMARY:
Dendrogenin A is present in mammals normal tissues and fluids, notably blood. It is down-represented or absent in cancer cell lines and tumors. In the opposite, OCDO is accumulated in cancerous conditions and virtually absent of normal tissues. This study will try to determine modulations of these oxysterols and protein involved in their metabolism between Acute myeloid leukemia (AML) patient samples and normal blood or marrow, for evaluation of these markers as companion biomarkers for Dendrogenin A treatment.

DETAILED DESCRIPTION:
Background : Acute myeloid leukemia is an unmet medical need since 5-year overall survival is 40-50% in younger adults and 10-15% in elderly. Dendrogenin A is a natural novel anticancer agent showing potent antileukemic activity which is under-represented in tumors. Dendrogenin A inhibits Cholesterol epoxide hydrolase and so modulates levels of substrates and products of this enzymatic complex.

Purpose : This is a biomedical study of interventional type which includes 30 patients and 30 blood samples as well as 5 marrow samples from healthy donors. It will last 24 month, 8 months recruiting and 16 months follow-up. Patients with acute myeloid leukemia for which an indication of chemotherapy treatment is retained will be enrolled in this study. This study will compare oxysterols (Dendrogenin A, 6-oxo-cholestane-3beta,5alpha-diol - OCDO) and related proteins as biomarkers of the disease between the two populations.

Interventions : The patients included in this study will be processed according to the standard treatment in force for their disease. This study does not in any way interfere with this treatment regimen, and is only based on additional samples of blood and bone marrow in acts planned in the prognostic or follow-up protocols. Treatment shall start within the 15 days following inclusion and first sampling.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of 18 years old or older
* Informed consent obtained and signed before any specific procedure in the study
* Patient member in a national insurance scheme

  * For patients with AML
* Men or women with a non promyelocytic acute myeloid leukemia as defined by WHO criteria and with at least 20% leukemic cells in blood at diagnosis
* for which treatment combining cytarabine and daunorubicin or idarubicin is retained
* WHO performance status ≤ 2

  * for healthy volunteers Criteria of eligibility for blood or bone marrow donation according to French Blood Institution

Exclusion criteria:

* Pregnant women or nursing mothers cannot participate in the study.
* Patients under legal guardianship.
* Any other medical or psychiatric condition or laboratory abnormality severe, acute or chronic making the inclusion of the patient in the study inappropriate in the opinion of the investigator.
* Patient unable to follow procedures, visits, examinations described in the study.

  * For patients with AML :
* Patients having received any anti-AML treatment with the exception of oral hydroxyurea.
* Patients for which a treatment different from the combination cytarabine+anthracycline has been selected

  * For healthy volunteers
* Criteria of ineligibility for blood donation according to EFS (French Blood Institution)
* For bone marrow : heart disease, high blood pressure, respiratory diseases, diseases of the nervous system history of cancers, diseases metabolic (diabetes, liver failure), history of recurring phlebitis or pulmonary embolism, disabling lumbar problems, neuromuscular diseases, angioedema, significant overweight,.
* Any long term treatment, except contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Difference of dendrogenin A between patients and healthy donors | day 1
  Comparison of levels of Dendrogenin A, oxysterols and related proteins between healthy volunteers and AML patients

SECONDARY OUTCOMES:
50 percent inhibitory concentration | day 1
  50 percent inhibitory concentration (evaluated by the rate of dead cells determined by a staining exclusion test and / or by flow cytometry) to assess the in vitro efficacy of Dendrogenin A in AML samples.

CONTACTS AND LOCATIONS:
Overall Officials: Christian RECHER, Doctor, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Chu Toulouse, Toulouse, France